CLINICAL TRIAL: NCT06782191
Title: Temporomandibular Joint Arthroscopic Lysis and Lavage Compared to Operative Arthroscopy in Disc Displacement With Reduction: a Randomised, Double-blind, Controlled Trial
Brief Title: TMJ Arthroscopic Lysis and Lavage Compared to Operative Arthroscopy in Disc Displacement With Reduction.
Acronym: ALLOAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Eastmaninstitutet (Other)
Responsible Party: Principal Investigator, Mattias Ulmner, Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-06478-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Joint Disc Displacement, With Reduction; Temporomandibular Disorders (TMD)
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic lysis and lavage (Active Comparator): Arthroscopic lysis and lavage refers to an arthroscopic procedure where the temporomandibular joint is rinsed with saline solution and where the joint capsule is distended and where adhesions are lysated bluntly. This is mananged through one port of entry into the joint.
  Interventions: Procedure: Arthroscopic lysis and lavage
- Operative arthroscopy (Experimental): Operative arthroscopy refers to an arthroscopic procedure where the temporomandibular joint is accessed via two ports of entry. The joint is rinsed with saline solution and the anterior disc attachment is released with cold ablation where after the posterior attachment is sclerosed with the coagulation mode on the coblator.
  Interventions: Procedure: Operative arthroscopy

INTERVENTIONS:
Procedure: Arthroscopic lysis and lavage — Arthroscopic lysis and lavage refers to an arthroscopic procedure where the temporomandibular joint is rinsed with saline solution and where the joint capsule is distended and where adhesions are lysated bluntly.
  Arms: Arthroscopic lysis and lavage
Procedure: Operative arthroscopy — Operative arthroscopy refers to an arthroscopic procedure where the temporomandibular joint is accessed via two ports of entry. The joint is rinsed with saline solution and the anterior disc attachment is released with cold ablation where after the posterior attachment is sclerosed with the coagulation mode on the coblator.
  Arms: Operative arthroscopy

SUMMARY:
The goal of this clinical trial is to compare the intervention arthroscopic lysis and lavage to the intervention operative arthroscopy in treating disabling and painful temporomandibular joint disc displacement with reduction. The main questions it aims to answer are:

* Which surgical method that best improves mouth opening capacity, TMJ pain, and TMJ disability?
* If any pre- or peri-operative variable/-s could be identified as a predictor for surgical outcome? Researchers will compare arthroscopic lysis and lavage to operative arthroscopy to see if operative arthroscopy works better to treat temporomandibular joint disc displacement.

Participants will:

* Have one of the two interventions under general anesthesia, not knowing which intervention.
* Visit an external clinic for regular checkups at 1, 3, 6, 12, and 24 months after surgery.
* Answer three different quality of life surveys at the checkups.

DETAILED DESCRIPTION:
1. BACKGROUND The temporomandibular joint (TMJ) is a bilateral joint comprised of two cartilage covered bone surfaces that articulates against each other during mouth opening and closing. A dense cartilage disc is situated between the two joint surfaces creating two separate joint compartments.

   Disc displacement (DD) is characterised by an improper position of the TMJ disc relative to the articulating surfaces and affects up to 30% of the population. DD with reduction (DDwR) is a sub-diagnosis of DD where the disc has got displaced, often in an anteromedial direction. During mouth opening the disc reduces into its right position with a snapping sound and on mouth closing the disc dislocates again. DDwR is often not affecting the patient but under somewhat unclear circumstances it might sometimes create pain and severe functional disability. A recent Swedish publication has shown that patients with TMJ disorders had significantly more days of work disability (2-3 times more) compared to a non-TMD cohort followed over a ten year period. The reliance on social security benefits in the group of patients that had TMJ surgery more than once were more accentuated compared to other TMJ disorder patients.

   The primary treatment for DDwR is non-surgical, most often physiotherapy and/or occlusal splint therapy. If non-surgical treatment fails the Swedish National Board of Health and Welfare primarily recommends open joint surgery, discectomy. TMJ arthroscopy in this situation has been assessed with a low level of evidence, thus not primarily recommended. Although, there are several publications rating arthroscopy as a potentially good DDwR treatment, but these publications often present their results mixing several TMJ diagnoses and most often in the form of retrospective case series, making clear conclusions hard to make. Another problem with present studies on TMJ arthroscopy due to DDwR is that successful treatment seldom is predefined as parameters to be fulfilled considering both clinical measurements and patient reported outcome. Instead, one parameter after another is analysed in singularity, which unfortunately do not give the reader the whole picture. Although, in a couple of studies a weighted success rate is demonstrated where arthroscopy seems very successful treating DDwR with rates between 81-90 %. This is well in parity with earlier studies on discectomy declaring around 85% success rate.When comparing the two different surgical methods discectomy and arthroscopy, arthroscopy is less invasive, almost no negative side effects, shorter operating time, and shorter rehabilitation and sick-leave.

   Arthroscopic treatment of DDwR has been described with two different methods, arthroscopic lysis and lavage (ALL) and operative arthroscopy with anterior release (OAA), never compared with each other in a randomised controlled fashion. ALL is performed with a rod-shaped lens inserted into the TMJ cavity enabling direct visualisation, The operative procedure involves manipulation of disc position, semi-blind release of adhesions (lysis), and irrigation (lavage) of the joint with either saline solution or Ringer's solution. Generally the procedure is performed under general anaesthesia, but there are reports on ALL performed in local anaesthesia or conscious sedation. OAA is basically an ALL expanded with an extra instrument canal/working cannula inserted into the TMJ enabling ablation of the anterior disc attachment and scarification (coagulation) of the posterior attachment under direct visualisation. The OAA procedure is performed under general anaesthesia. Comparing ALL and OAA has been done in a retrospective manner, and in patients with DDwR there were a 30% difference in MIO postoperative at 6 months in favour of OAA and almost the same difference when considering TMJ pain.

   Synovial fluid from the TMJ has been used since the mid-90's mostly for analysing inflammatory markers. Proteomics is a relatively new technique for analysing protein profiles and has only been applied a couple of times in the field of TMJ pathology. Since the aetiology of DD is still not known, proteomics provides a comprehensive insight of the protein profile of TMJ disorders.

   There are no RCT's comparing the outcome of ALL and OAA in patients with DDwR. The aim of this study is to evaluate outcome of ALL and OAA in treating DDwR in a double-blind fashion. A secondary aim is to describe the protein profile in patients with DDR and to see if patient-specific differences might be connected to surgical outcome, local inflammation, or local pain.
2. HYPOTHESIS/RESEARCH QUESTIONS OAA has a superior outcome compared to ALL treating patients with DDwR. The outcome will be longitudinally evaluated with a combination of maximum mouth opening capacity, patient reported TMJ pain and TMJ disability, and Quality of life (QoL) questionnaires at pre-determined time-points during a 24-month postoperative period.

   The primary research question is which of the two surgical methods that best improves the above stated variables.

   Secondary questions are:
   * Is there an identifiable protein profile regarding DDwR.
   * could any pre- or peri-operative variable/-s be identified as a predictor for outcome.
   * what is the impact from DDwR on QoL and the surgical outcomes impact on QoL.
   * are there any differences in how fast the patient recover after ALL and OAA, respectively.
   * has the discs position been altered due to applied surgical intervention.
   * can the patient-reported variable "TMJ disability" work as a possible substitute for JFSL-8.
3. METHODS 3.1. Study design

Randomised, double-blind, controlled trial where the outcome of ALL and OAA treatment due to DDwR is compared.

3.2. Data source

All patients referred to the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, with the diagnosis DDwR and with a history of not responding to non-surgical treatment will be screened for inclusion.

3.3 Exposure/Intervention

Patients will be randomly assigned to either ALL or OAA. Both treatments will be performed under general anaesthesia. The randomisation will be made in blocks of two in a 1:1 ratio. A computer software provided by KTA (Karolinska Trial Alliance) will handle the randomisation process. At time of surgery, when the patient is under general anaesthesia and draped in sterile cloth, the patient will be allocated to either ALL or OAA. In this manner the intervention or placebo treatment will be blinded to the patient but not to the surgeon. The person evaluating the outcome of surgery (the assessor) will not know which treatment the patient has undertaken. The two surgical procedures are described below.

ALL: The surgical procedure is performed according to the original description of the technique. During the operation the joint space is irrigated with a minimum of 300 mL saline solution. A pressure infuser (InfuseITTM) set at 175 mmHg will be used to standardise the irrigation pressure. At the start of joint irrigation, the first 50 mL outflow irrigation fluid will be collected in a sterile container for later proteomic analysis. An extra stab incision will be performed approximately 2 cm ventral to the preauricular incision, in order to mimic an OAA intervention, please see below. At the end of surgery, the joint is flushed with 10 mL of Marcaine-Adrenaline (5.0 mg/mL). No other medication will be injected or otherwise introduced into the joint compartment. The incisions are sutured with a single non-resorbable suture, and a wound dressing is put over the incision. The described intervention is standardized and takes 20-30 minutes.

OAA: a description of the technique was made by McCain et al. The operation follows the steps of ALL, but adds instrumentation (coblation probe, Reflex Ultra 45, ArthroCare) of the joint under direct visualisation. An anterolateral release of the disc attachment is performed, the disc is mobilised with the blunt obturator, and a scarification/coagulation of the posterior ligament is performed with the coblation probe. During the operation the joint space is irrigated with a minimum of 300 mL saline solution. A pressure infuser (InfuseITTM) set at 175 mmHg will be used to standardise the irrigation pressure. At the start of joint irrigation, the first 50 mL outflow irrigation fluid will be collected in a sterile container for later proteomics. Finally, the joint is flushed with 10 mL of Marcaine-Adrenalin (5.0 mg/mL) and the incisions sutured with a single non-resorbable suture each. The intervention takes 30-40 minutes.

To keep the blinding intact for the patient and the assessor, the medical chart will be written as if all the patients had ALL performed.

Both the intervention groups will have postoperative physiotherapy training for a period of one month from the day after surgery in accordance with a specified home exercise program (see attachment). If needed, the home exercise program can be prolonged or individually adjusted after the first month for up to an additional month. If the patient uses an occlusal splint prior to surgery the splint may have to be adjusted and that has to be performed by the assessor.

After approximately 6 months postoperatively an MRI will be performed to monitor the discs position.

3.4. Outcome

Please, see "Outcome measures" below.

3.5. Sample size

48 patients in each intervention group, i.e. 96 patients in total, in accordance with the power analysis, see "Statistical analysis".

3.6. Inclusion and exclusion criteria

Please, see "Eligibility" below.

3.7. Data collection

At registration for surgery and after obtained informed consent, baseline data is collected by the surgeon designating the patient to surgery (see attachment). Predetermined follow-up visits are at 1 week when the surgeon will remove the stich and do a reinstruction for the home-exercise program, and at 1, 3, 6, 12, and 24 months postoperative when the assessor examine the patient according to the specific exam protocol (see attachment). The assessor/-s will be calibrated alongside the surgeon/-s before the start of the study in accordance with the DC/TMD criteria. At 6-month intervals the surgeons and assessors will have a meeting for re-calibrating purposes. To determine any change in disc position an MRI will be performed approximately 6 months postoperative.

Objective data only registered preoperative: name, personal identification number, age, sex, affected joint (left, right).

Objective data registered both pre- and post-operatively: MIO with and without pain (mm), lateral excursive movement (mm), protrusion (mm), pain upon palpating masticatory muscles, pain upon lateral joint palpation.

Subjective data registered both pre- and post-operatively: patient-reported TMJ disability (NRS 0-10), patient-reported TMJ pain (NRS 0-10), patient-reported psycho-social impairment because of TMJ disorder (NRS 0-10), patient-reported global pain (NRS 0-10), and quality of life questionnaire EQ-5D-5L, JFSL-8, and OHIP 14-S.

Perioperative data: antibiotic prophylaxis (yes/no), performed surgery (ALL/OAA), maximum assisted mouth opening (mm), duration of surgery (min), duration of general anaesthesia (min), lavage volume (mL), preauricular swelling due to lavage (yes/no), negative event during and due to surgery. Grading of intraarticular conditions will be made according to the scale proposed by Gynther et al.: synovitis (0-3), degenerative changes (0-3), and fibrosis/adhesions (0-2).[36, 37]

3.8 Revelation of blinding

At the 6-month visit the patients will be asked if they believe that they had ALL or OAA. The assessor will also give their opinion in that matter. After the 6-month follow-up, the blinding will be revealed to the patient if they want to. Patients with a non-successful outcome might be offered another therapy; non-surgical or surgical. Controls will be made at 12- and 24-months post-operative regarding all patients. Additional information about the surgical intervention (OAA) will be added to the affected patients' medical record.

3.9. Analysis of synovial fluid Proteomic analysis and protein quantification in synovial fluid will be performed at PainOmics laboratory, University hospital in Linköping. In this project, we will follow a discover and verification/validation schema. In the first step peptides and protein contents of the synovial fluid will be analysed using 2-DE in combination with mass spectrometry. With this technique it is possible to separate and quantify more than 1000 proteins and it is the only technique that allows separating and studying different protein isoforms. Quantification of the separated proteins is achieved by spot integration using specialized 2-DE software that makes it possible to compare protein patterns from different subjects/groups. Identification of the protein is performed by in-gel digestion of each protein, recovery of the fragments from the gel, and analysis by mass spectrometry (MS) using MALDI-T.

4. STATISTICAL ANALYSIS The primary objective is to evaluate the superiority of OAA compared to ALL in patients diagnosed with DDwR and not responding to non-surgical treatment. The outcome variable is dichotomous (successful/not successful) where a successful outcome in the OAA group is assessed to be 89 % and in the ALL group 64 %. With 80 % power and a 5 % significance level the groups must contain 44 patients each. Dropout rate of 10 % is accounted for which means that 48 patients/group must be included to verify superiority.

Statistical analyses will be performed using the Chi-Square test for bivariate data and the Students t-test (unpaired and paired) for mean values, as well as repeated measures ANOVA. Longitudinal data will be analysed with linear regression analysis and predictors for surgical outcome will be evaluated through logistic regression. The intention to treat analysis model will be used.

Potential known confounders may be adjusted for in the analysis and the risk of residual unknown confounders should be reduced by the randomisation process.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral DDwR verified with clinical and magnetic resonance imaging (MRI) findings
* TMJ pain ≥ 3 (NRS) and/or TMJ disability ≥ 3 (NRS)
* Age ≥ 18 years

Exclusion Criteria:

* Prior open TMJ surgery
* Patient diagnosed with rheumatologic joint disease
* ASA (American Society of Anaesthesiologists) > 3
* Patient unable to verify informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome | From intervention to the 6 month postoperative follow up.
  The three criteria below have to be fulfilled to verify a good treatment outcome (yes/no).
  1. Maximum interincisal opening (MIO) of ≥ 35 mm, or an increase of MIO of ≥ 40 %.
  2. Patient-reported TMJ pain. Visual analogue scale (VAS) ≤ 3, or ≤ 40% reduction.
  3. Patient-reported TMJ disability. VAS ≤ 3, or a 40 % reduction.

SECONDARY OUTCOMES:
Qulity of life surveys | From intervention to the 6 month postoperative follow up.
  To evaluate EQ-5D-5L, JFSL-8, and OHIP 14-S and what impact DDwR has got on QoL and difference in QoL after interventions,

OTHER OUTCOMES:
Pain in the temporomandibular joint (TMJ) during function | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate how much pain TMJ function (opening, biting, chewing, speaking, etc.) has caused on average over the past 2-week period. This estimation should exclude the worst imaginable pain. Each TMJ is assessed individually, meaning the patient should provide a numerical value between 0 (no pain) and 10 (worst imaginable pain) for each joint.
Pain in the temporomandibular joint at rest | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate pain in each TMJ at rest on a scale graded from 0 to 10. The value should reflect an average representative of the past 2-week period.
Functional impairment of the temporomandibular joint | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the degree of functional impairment caused by current TMJ issues. This variable includes both joint mobility and the ability to consume food. The scale is graded from 0 to 10. A score of 0 indicates no impairment, meaning unrestricted jaw opening and the ability to eat all types of food without difficulty. A score of 10 represents complete functional impairment, such as zero millimeters of opening or being able to consume only liquids due to the inability to chew solid food.
Psychosocial impact | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the psychosocial impact of their TMJ issues from 0 to 10. A score of 0 indicates no impact, while a score of 10 represents the worst imaginable impact. This may include how much and how often the patient thinks about their TMJ issues, how it affects their mood, and how it impacts their social life, such as withdrawing from social interactions.
Other bodily pain | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the degree of bodily pain unrelated to TMJ pain between 0 to 10. This can include pain from other joints, gastrointestinal discomfort, etc. A score of 0 indicates no other bodily pain, while a score of 10 indicates the worst imaginable bodily pain.
Palpation tenderness of TMJ | From intervention to the 6 month postoperative follow up.
  The TMJ is palpated laterally according to DC/TMD (500 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Palpation tenderness of the masseter and temporalis muscles: | From intervention to the 6 month postoperative follow up.
  The masseter and temporalis muscles are palpated at three separate sites each, according to DC/TMD (1000 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Maximum interincisal opening | From intervention to the 6 month postoperative follow up.
  Measured in millimeters. The distance between teeth 11 and 41 is measured as the patient opens their mouth as wide as possible. If this is not feasible due to malocclusion, tooth loss, etc., an alternative representative pair of front teeth is chosen for measurement. This should be noted in the patient's record to ensure consistent measurements in the future.
Maximum protrusion | From intervention to the 10 year follow up.
  Horizontal overbite (HOB) is first measured in millimeters during habitual intercuspal position. The value is positive if tooth 11 is located facially to tooth 41 and negative if the reverse is true. The patient is then instructed to protrude the mandible maximally, and the horizontal distance between the incisal edges of teeth 11 and 41 is measured again. These two measurements are then added together (noting negative HOB in Class III cases).
Maximum laterotrusion | From intervention to the 6 month postoperative follow up.
  The patient is instructed to move the mandible to one side. The distance between the midline of the maxilla (between teeth 11 and 21) and the midline of the mandible (between teeth 31 and 41) is measured in millimeters. Any midline deviation during habitual intercuspal position is measured and subtracted from or added to the recorded value. Laterotrusion is measured for both left and right movements.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ulmner, DDS, PhD, Principal Investigator — Karolinska Institutet, Department of Dental Medicine
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP is available through ClinicalTrials.

REFERENCES:
- [Background] Wilkes CH. Internal derangements of the temporomandibular joint. Pathological variations. Arch Otolaryngol Head Neck Surg. 1989 Apr;115(4):469-77. doi: 10.1001/archotol.1989.01860280067019. PMID 2923691
- [Background] Wieckiewicz M, Boening K, Wiland P, Shiau YY, Paradowska-Stolarz A. Reported concepts for the treatment modalities and pain management of temporomandibular disorders. J Headache Pain. 2015;16:106. doi: 10.1186/s10194-015-0586-5. Epub 2015 Dec 7. PMID 26644030
- [Background] Ulmner M, Sugars R, Naimi-Akbar A, Alstergren P, Lund B. Cytokines in temporomandibular joint synovial fluid and tissue in relation to inflammation. J Oral Rehabil. 2022 Jun;49(6):599-607. doi: 10.1111/joor.13321. Epub 2022 Apr 9. PMID 35342975
- [Background] Ulmner M, Kruger-Weiner C, Lund B. Patient-Specific Factors Predicting Outcome of Temporomandibular Joint Arthroscopy: A 6-Year Retrospective Study. J Oral Maxillofac Surg. 2017 Aug;75(8):1643.e1-1643.e7. doi: 10.1016/j.joms.2017.04.005. Epub 2017 Apr 13. PMID 28487216
- [Background] Smolka W, Yanai C, Smolka K, Iizuka T. Efficiency of arthroscopic lysis and lavage for internal derangement of the temporomandibular joint correlated with Wilkes classification. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Sep;106(3):317-23. doi: 10.1016/j.tripleo.2007.12.007. Epub 2008 Jan 15. PMID 18226569
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Sanders B. Arthroscopic surgery of the temporomandibular joint: treatment of internal derangement with persistent closed lock. Oral Surg Oral Med Oral Pathol. 1986 Oct;62(4):361-72. doi: 10.1016/0030-4220(86)90282-3. PMID 3464910
- [Background] Salinas Fredricson A, Kruger Weiner C, Adami J, Rosen A, Lund B, Hedenberg-Magnusson B, Fredriksson L, Svedberg P, Naimi-Akbar A. Sick leave and disability pension in a cohort of TMD-patients - The Swedish National Registry Studies for Surgically Treated TMD (SWEREG-TMD). BMC Public Health. 2022 May 9;22(1):916. doi: 10.1186/s12889-022-13329-z. PMID 35534826
- [Background] Sale H, Bryndahl F, Isberg A. Temporomandibular joints in asymptomatic and symptomatic nonpatient volunteers: a prospective 15-year follow-up clinical and MR imaging study. Radiology. 2013 Apr;267(1):183-94. doi: 10.1148/radiol.12112243. Epub 2012 Dec 18. PMID 23249569
- [Background] Nyberg J, Adell R, Svensson B. Temporomandibular joint discectomy for treatment of unilateral internal derangements--a 5 year follow-up evaluation. Int J Oral Maxillofac Surg. 2004 Jan;33(1):8-12. doi: 10.1054/ijom.2002.0453. PMID 14690653
- [Background] Miloro M, McKnight M, Han MD, Markiewicz MR. Discectomy without replacement improves function in patients with internal derangement of the temporomandibular joint. J Craniomaxillofac Surg. 2017 Sep;45(9):1425-1431. doi: 10.1016/j.jcms.2017.07.003. Epub 2017 Jul 17. PMID 28800843
- [Background] McCain JP, Sanders B, Koslin MG, Quinn JH, Peters PB, Indresano AT. Temporomandibular joint arthroscopy: a 6-year multicenter retrospective study of 4,831 joints. J Oral Maxillofac Surg. 1992 Sep;50(9):926-30. doi: 10.1016/0278-2391(92)90047-4. PMID 1506966
- [Background] McCain JP, de la Rua H, LeBlanc WG. Puncture technique and portals of entry for diagnostic and operative arthroscopy of the temporomandibular joint. Arthroscopy. 1991;7(2):221-32. doi: 10.1016/0749-8063(91)90111-a. PMID 2069635
- [Background] Liu X, Yang Y, Chen L, Tian S, Abdelrehem A, Feng J, Fu G, Chen W, Ding C, Luo Y, Zou D, Yang C. Proteome Analysis of Temporomandibular Joint with Disc Displacement. J Dent Res. 2022 Dec;101(13):1580-1589. doi: 10.1177/00220345221110099. Epub 2022 Oct 20. PMID 36267015
- [Background] Kellesarian SV, Al-Kheraif AA, Vohra F, Ghanem A, Malmstrom H, Romanos GE, Javed F. Cytokine profile in the synovial fluid of patients with temporomandibular joint disorders: A systematic review. Cytokine. 2016 Jan;77:98-106. doi: 10.1016/j.cyto.2015.11.005. Epub 2015 Nov 7. PMID 26556103
- [Background] Kaneyama K, Segami N, Sun W, Sato J, Fujimura K. Analysis of tumor necrosis factor-alpha, interleukin-6, interleukin-1beta, soluble tumor necrosis factor receptors I and II, interleukin-6 soluble receptor, interleukin-1 soluble receptor type II, interleukin-1 receptor antagonist, and protein in the synovial fluid of patients with temporomandibular joint disorders. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Mar;99(3):276-84. doi: 10.1016/j.tripleo.2004.06.074. PMID 15716832
- [Background] Kaneyama K, Segami N, Sato J, Murakami K, Iizuka T. Outcomes of 152 temporomandibular joints following arthroscopic anterolateral capsular release by holmium: YAG laser or electrocautery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 May;97(5):546-51; discussion 552. doi: 10.1016/S1079210403007261. PMID 15153864
- [Background] Jasim H, Ernberg M, Carlsson A, Gerdle B, Ghafouri B. Protein Signature in Saliva of Temporomandibular Disorders Myalgia. Int J Mol Sci. 2020 Apr 7;21(7):2569. doi: 10.3390/ijms21072569. PMID 32272779
- [Background] Holmlund AB, Gynther G, Axelsson S. Diskectomy in treatment of internal derangement of the temporomandibular joint. Follow-up at 1, 3, and 5 years. Oral Surg Oral Med Oral Pathol. 1993 Sep;76(3):266-71. doi: 10.1016/0030-4220(93)90250-8. PMID 8378038
- [Background] Holmlund AB, Axelsson S, Gynther GW. A comparison of discectomy and arthroscopic lysis and lavage for the treatment of chronic closed lock of the temporomandibular joint: a randomized outcome study. J Oral Maxillofac Surg. 2001 Sep;59(9):972-7; discussion 977-8. doi: 10.1053/joms.2001.25818. PMID 11526556
- [Background] Holmlund A, Gynther G, Axelsson S. Efficacy of arthroscopic lysis and lavage in patients with chronic locking of the temporomandibular joint. Int J Oral Maxillofac Surg. 1994 Oct;23(5):262-5. doi: 10.1016/s0901-5027(05)80104-3. PMID 7890964
- [Background] Herr MM, Fries KM, Upton LG, Edsberg LE. Potential biomarkers of temporomandibular joint disorders. J Oral Maxillofac Surg. 2011 Jan;69(1):41-7. doi: 10.1016/j.joms.2010.05.013. PMID 21163381
- [Background] Gynther GW, Holmlund AB, Reinholt FP, Lindblad S. Temporomandibular joint involvement in generalized osteoarthritis and rheumatoid arthritis: a clinical, arthroscopic, histologic, and immunohistochemical study. Int J Oral Maxillofac Surg. 1997 Feb;26(1):10-6. doi: 10.1016/s0901-5027(97)80838-7. PMID 9081245
- [Background] Gynther GW, Holmlund AB, Reinholt FP. Synovitis in internal derangement of the temporomandibular joint: correlation between arthroscopic and histologic findings. J Oral Maxillofac Surg. 1994 Sep;52(9):913-7; discussion 918. doi: 10.1016/s0278-2391(10)80066-7. PMID 8064453
- [Background] Gonzalez-Garcia R, Rodriguez-Campo FJ, Escorial-Hernandez V, Munoz-Guerra MF, Sastre-Perez J, Naval-Gias L, Gil-Diez Usandizaga JL. Complications of temporomandibular joint arthroscopy: a retrospective analytic study of 670 arthroscopic procedures. J Oral Maxillofac Surg. 2006 Nov;64(11):1587-91. doi: 10.1016/j.joms.2005.12.058. PMID 17052583
- [Background] Gonzalez-Garcia R, Rodriguez-Campo FJ. Arthroscopic lysis and lavage versus operative arthroscopy in the outcome of temporomandibular joint internal derangement: a comparative study based on Wilkes stages. J Oral Maxillofac Surg. 2011 Oct;69(10):2513-24. doi: 10.1016/j.joms.2011.05.027. PMID 21939814
- [Background] Gonzalez LV, Lopez JP, Diaz-Baez D, Orjuela MP, Chavez M. Clinical outcomes of operative arthroscopy and temporomandibular medical infiltration with platelet-rich fibrin in upper and lower articular space. J Craniomaxillofac Surg. 2021 Dec;49(12):1162-1168. doi: 10.1016/j.jcms.2021.07.001. Epub 2021 Aug 3. PMID 34384651
- [Background] Fu K, Ma X, Zhang Z, Chen W. Tumor necrosis factor in synovial fluid of patients with temporomandibular disorders. J Oral Maxillofac Surg. 1995 Apr;53(4):424-6. doi: 10.1016/0278-2391(95)90717-3. PMID 7699497
- [Background] Fernandez Sanroman J, Costas Lopez A, Fernandez Ferro M, de Sanchez AL, Stavaru B, Arenaz Bua J. Complications of temporomandibular joint arthroscopy using two-portal coblation technologies: A prospective study of 475 procedures. J Craniomaxillofac Surg. 2016 Sep;44(9):1221-5. doi: 10.1016/j.jcms.2016.06.027. Epub 2016 Jul 2. PMID 27443801
- [Background] Eriksson L, Westesson PL. Discectomy as an effective treatment for painful temporomandibular joint internal derangement: a 5-year clinical and radiographic follow-up. J Oral Maxillofac Surg. 2001 Jul;59(7):750-8; discussion 758-9. doi: 10.1053/joms.2001.24288. PMID 11429734
- [Background] Doetzer AD, Herai RH, Buzalaf MAR, Trevilatto PC. Proteomic Expression Profile in Human Temporomandibular Joint Dysfunction. Diagnostics (Basel). 2021 Mar 28;11(4):601. doi: 10.3390/diagnostics11040601. PMID 33800589
- [Background] Chowdhury SKR, Saxena V, Rajkumar K, Shadamarshan RA. Complications of Diagnostic TMJ Arthroscopy: An Institutional Study. J Maxillofac Oral Surg. 2019 Dec;18(4):531-535. doi: 10.1007/s12663-019-01202-3. Epub 2019 Feb 26. PMID 31624430
- [Background] Chossegros C, Cheynet F, Gola R, Pauzie F, Arnaud R, Blanc JL. Clinical results of therapeutic temporomandibular joint arthroscopy: a prospective study of 34 arthroscopies with prediscal section and retrodiscal coagulation. Br J Oral Maxillofac Surg. 1996 Dec;34(6):504-7. doi: 10.1016/s0266-4356(96)90245-4. PMID 8971443
- [Background] Bjornland T, Larheim TA. Discectomy of the temporomandibular joint: 3-year follow-up as a predictor of the 10-year outcome. J Oral Maxillofac Surg. 2003 Jan;61(1):55-60. doi: 10.1053/joms.2003.50010. PMID 12524609
- [Background] Al-Baghdadi M, Durham J, Steele J. Timing interventions in relation to temporomandibular joint closed lock duration: a systematic review of 'locking duration'. J Oral Rehabil. 2014 Jan;41(1):24-58. doi: 10.1111/joor.12126. Epub 2014 Jan 7. PMID 24393132
- [Background] Abboud W, Yahalom R, Givol N. Treatment of Intermittent Locking of the Jaw in Wilkes Stage II Derangement by Arthroscopic Lysis and Lavage. J Oral Maxillofac Surg. 2015 Aug;73(8):1466-72. doi: 10.1016/j.joms.2015.02.027. Epub 2015 Mar 18. PMID 25970513